CLINICAL TRIAL: NCT01072708
Title: Determination of the Predictive Factors in the Reversibility or the Aggravation in the Disorders of the Glucose Metabolism in Cystic Fibrosis Patients (Study DIAMUCO)
Brief Title: Determination of the Predictive Factors in the Reversibility or the Aggravation in the Disorders of the Glucose Metabolism in Cystic Fibrosis Patients
Acronym: DIAMUCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2008.523/24
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Diabetes in Cystic Fibrosis Patients
Keywords: Cystic fibrosis -diabetes - glucose tolerance - reversibility - oral glucose tolerance test - predictive factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Prospective cohort with an annual follow-up — Annualfollow-up including :
  * oral glucose tolerance test
  * dietary survey
  * biological evaluation
  * bacteriological and respiratory measures
  * dual-energy x-ray absorptiometry
  * physical activity survey

SUMMARY:
For some years, the investigators observe an increase of the arisen of diabetes in cystic fibrosis patients However, this diabetes may be reversible. The investigators speak about " Cystic fibrosis related diabetes.". The objective of this project, is to know better what facilitates the appearance and the reversibility of the diabetes, such as the genetic mutations, the respiratory state and the lung infections. Theses knowledges should allow to adapt the screening of diabetes, and its treatment, for the patients affected by cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patients with at least one visit in Cystic fibrosis Center in Rhône-Alpes (France) during the second half-year 2008
* Patients with disorders or not of the glucose metabolism
* Patient with pancreatic insufficiency

Exclusion Criteria:

* Patient with hypoglycemia treatment : insulin or oral antidiabetic
* Patient with an age < 10 years
* Patient with lung transplant

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Describe the natural history of the glucose tolerance in cystic fibrosis patients and to identify the predictive factors of the reversibility or the aggravation in the disorders of the glucidic metabolism. | 3 years

SECONDARY OUTCOMES:
Estimate prevalence of the various stages of disorders of the glucose metabolism : glucose intolerance and diabetes | 3 years
Estimate the probability of arisen the complications associated to the disorders of the glucidic metabolism : - deterioration of the respiratory function, - lung exacerbations - alteration of the nutritional state | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Interne - Centre Hospitalier Lyon Sud, Pierre-Bénite, France

REFERENCES:
- [Background] Reynaud Q, Rabilloud M, Roche S, Poupon-Bourdy S, Iwaz J, Nove-Josserand R, Blond E, Laville M, Llerena C, Quetant S, Reix P, Touzet S, Durieu I. Glucose trajectories in cystic fibrosis and their association with pulmonary function. J Cyst Fibros. 2018 May;17(3):400-406. doi: 10.1016/j.jcf.2017.09.010. Epub 2017 Oct 14. PMID 29037538